CLINICAL TRIAL: NCT01351714
Title: Safe D3 Right Hemicolectomy for Cancer Through 3D MDCT Angiography Reconstruction
Brief Title: Safe D3 Right Hemicolectomy for Cancer Through Multidetector Computed Tomography (MDCT) Angio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Konya Meram State Hospital (Other); University of Geneva, Switzerland (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Dejan Ignjatovic, MD, PhD, Professor, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3 MDCT angio
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Colon Cancer
Keywords: D3 resection; right colectomy; MDCT angiography; lymphadenectomy; safe; right colon; preoperative
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- D3 resection (Other): Radical D3 resection of the right colon through the use of preoperative MDCT angiography
  Interventions: Procedure: D3 resection

INTERVENTIONS:
Procedure: D3 resection — Radical D3 resection of the right colon through the use of preoperative MDCT angiography

SUMMARY:
When performing a resection of the right colon due to cancer one aims not only to remove the tumor bearing bowel segment, but also lymph nodes draining the affected area. These lymph nodes are located along the arteries supplying the right colon. Through using a preoperative CT scan which can map these arteries very precisely one can ligate these vessels closer to their origin and thus remove more lymph nodes which may potentially harbor cancer cells. This study aims to compare patients operated more radically through use of preoperative CT which maps the mentioned arteries with patients operated in the standard way.

DETAILED DESCRIPTION:
The Norwegian gastrointestinal cancer group has recommended D3 resection as the standard operative technique for colon cancer. D3 resection implies ligation of the blood vessels at their origin. There is evidence that the recurrence free period and survival improves with the number of lymph nodes harvested at surgery. However, the current practice in Norway, while performing right hemicolectomy for cancer is to ligate the feeding vessels for the right colon on the right hand side of the superior mesenteric vein (SMV). Significant arterial stumps have been demonstrated in patients operated for right colon cancer with this technique (right colic artery and ileocolic artery vascular stumps with an average length of 3.5 cm and 2.5 cm, respectively). This leaves reason to believe that a certain number of central lymph nodes remain after the procedure.

The complex anatomical relationship between the right colic artery and ileocolic artery with the superior mesenteric vein make D3 resection demanding, especially if the right colic artery lies posterior to the SMV. These relationships are investigated in detail in postmortem anatomical studies. These studies show that the right colic artery lies most often anterior to the SMV, while the ileocolic artery lies most often posterior to the SMV. Data has also been provided that a CT angiography can verify these relations as well as postmortem anatomical studies in living patients, thus allowing the surgeon to be aware of them prior to surgery. This could prove to be crucial in planning the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histo-pathologically verified adeno-carcinoma of the right colon
* Patients under the age of 75
* Patients medically cleared by anesthesiologist for general anesthesia
* Signed informed consent form

Exclusion Criteria:

* Patients with recurrent cancer after previous surgery
* Patients with distant metastasis
* Patients who are not medically cleared to undergo anesthesia
* Patients who do not sign the informed consent form

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2011-05; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Number of additional lymph nodes removed through radical D3 resection | 1 year
  The short term outcome of this study will compare number of lymph nodes removed, operating time and complications between the two groups.

SECONDARY OUTCOMES:
Disease free survival 2 and 5 years after initial surgery | 5 years
  One will compare disease free survival at 2 and 5 years between the two groups to see if those more radically operated through D3 resection will have better outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lorenskog
  - Vestfold Hospital Trust, Tønsberg

REFERENCES:
- [Derived] Banipal GS, Stimec BV, Andersen SN, Faerden AE, Edwin B, Baral J, Nesgaard JM, Benth JS, Ignjatovic D; R. C. C. study group. Comparing 5-Year Survival Rates Before and After Re-stratification of Stage I-III Right-Sided Colon Cancer Patients by Establishing the Presence/Absence of Occult Tumor Cells and Lymph Node Metastases in the Different Levels of Surgical Dissection. J Gastrointest Surg. 2022 Oct;26(10):2201-2211. doi: 10.1007/s11605-022-05434-6. Epub 2022 Aug 29. PMID 36036877
- [Derived] Banipal GS, Stimec BV, Andersen SN, Faerden AE, Edwin B, Baral J, Benth JS, Ignjatovic D; RCC study group. Interactions of occult tumor spread and surgical technique on overall and disease-free survival in patients operated for stage I and II right-sided colon cancer. J Cancer Res Clin Oncol. 2021 Dec;147(12):3535-3543. doi: 10.1007/s00432-021-03773-6. Epub 2021 Aug 24. PMID 34427788